CLINICAL TRIAL: NCT00151580
Title: Comparison of Maintenance Treatment by Ribavirin to a Placebo, After an Initial One-year Treatment With Pegylated Interferon-α2a - Ribavirin Association in Hepatitis C Viral Recurrence After Liver Transplantation
Brief Title: Treatment of Recurrent Hepatitis C After Liver Transplantation
Acronym: TRANSPEG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government); ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: AFSSAPS 010588; PHRC/00-02; CIC0203/049
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2007-11

CONDITIONS: Liver Transplantation; Hepatitis C
Keywords: Hepatitis C; Viral recurrence; Ribavirin / Interferon
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Ribavirin maintenance treatment
  Interventions: Drug: Ribavirin
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ribavirin — 18 months of oral ribavirin maintenance treatment
  Arms: 1
Drug: Placebo — 18 months oral placebo treatment
  Arms: 2

SUMMARY:
In France, 50% of the hepatitis C virus carriers develop chronic clinical hepatitis, which may lead to cirrhosis and liver transplantation. Transplant infection by hepatitis C virus is constant after transplantation. This recurrence usually causes chronic liver disease, in 50 to 80% of the patients. The interest of a long-term treatment with ribavirin alone after transplantation has not been clearly demonstrated. The objective of our study is to evaluate the efficacy of ribavirin as a maintenance treatment after a one year interferon-α / ribavirin therapy on hepatitis C recurrence in the transplanted liver.

DETAILED DESCRIPTION:
Several therapeutic patterns have been described for the treatment of hepatitis C post-transplantation recurrence. A combination treatment associating interferon-α and ribavirin has shown some efficacy, but this efficacy has not been assessed yet in a placebo-controlled double-blind clinical trial. In our study, all included transplanted patients will be treated during 1 year with interferon-α and ribavirin. At the end of this period, they will be randomized to receive a maintenance treatment with ribavirin or a placebo for 1 additional year. Efficacy will be assessed on virological response after 30 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* First liver transplantation or retransplantation in the month after initial transplantation
* Patients aged over 18 years
* Post-hepatitis C cirrhosis
* Equilibrated immunosuppressive treatment
* Positive PCR for hepatitis C virus
* Liver biopsy between 6 months and 5 years after the transplantation with a fibrosis Metavir score at least F1
* Hemoglobin ≥ 10 g/dl
* Platelet count ≥ 50.000/mm3
* Normal TSH value
* Serum creatinine < 200µmol/l
* Informed written consent

Exclusion Criteria:

* Chronic rejection
* Acute rejection at inclusion
* Multi-visceral transplantation
* Renal or cardiac failure, severe sepsis
* Uncontrolled diabetes
* Positive serology for hepatitis B or HIV at inclusion
* EBV virus replication at inclusion
* Hepatocellular carcinoma at inclusion
* Cirrhosis with a fibrosis Metavir score F4 at inclusion
* Inclusion in another clinical trial less than one month ago
* Pregnancy
* Contra-indication to ribavirin or interferon
* History of or current psychiatric troubles
* Thyroid disease uncontrolled by treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2002-02; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Negative viral PCR | 30 months

SECONDARY OUTCOMES:
Histological improvement | 30 months
Biological hepatic markers | 30 months
Quality of life | 30 months
Intensity, severity and delay to acute transplant rejection, histologically proven | 30 months
Incidence of death or graft loss | 30 months
Number of patients stopping the treatment and causes | 30 months
Incidence of adverse events classically related to treatment | 30 months
Incidence of adverse events possibly related to treatment | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Karim Boudjema, MD, PhD, Principal Investigator — CHU Rennes; Yvon Calmus, MD, Principal Investigator — AP-HP Hôpital Cochin
Locations (16):
- France (16):
  - Service d'Hépatologie - Hôpital Jean Minjoz, Besançon
  - Service de Chirurgie Digestive - Groupe Hospitalier Pellerin-Tripode, Bordeaux
  - Service d'Hépatogastroentérologie - Hôpital Beaujon, Clichy
  - Service d'Hépatologie et Gastroentérologie - Hôpital Henri Mondor, Créteil
  - Service des Maladies de l'Appareil Digestif - CHRU Claude Huriez, Lille
  - Médecine Digestive - Hôtel Dieu, Lyon
  - Service de Chirurgie Générale - Hôpital Edouard Herriot, Lyon
  - Chirurgie Générale - Hôpital de la Conception, Marseille
  - Service d'Hépaogastroentérologie - Hôpital Saint Eloi, Montpellier
  - Chirurgie Viscérale et Digestive -Hôpital de l'Archet, Nice
  - Service Hépato-gastroentérologie - Hôpital Saint Antoine, Paris
  - Service de Chirurgie Générale et Digestive - Hôpital Cochin, Paris
  - Département de Chirurgie Viscérale- Hôpital Pontchaillou, Rennes
  - Service de Chirurgie Générale et Transplantation Multi-organe - Hôpital de la Hautepierre, Strasbourg
  - Hôpital de Rangueil, Toulouse
  - Centre Hépato-biliaire - Hôpital Paul Brousse, Villejuif

REFERENCES:
- [Background] Cattral MS, Hemming AW, Wanless IR, Al Ashgar H, Krajden M, Lilly L, Greig PD, Levy GA. Outcome of long-term ribavirin therapy for recurrent hepatitis C after liver transplantation. Transplantation. 1999 May 15;67(9):1277-80. doi: 10.1097/00007890-199905150-00014. PMID 10342322
- [Background] Berenguer M, Prieto M, Cordoba J, Rayon JM, Carrasco D, Olaso V, San-Juan F, Gobernado M, Mir J, Berenguer J. Early development of chronic active hepatitis in recurrent hepatitis C virus infection after liver transplantation: association with treatment of rejection. J Hepatol. 1998 May;28(5):756-63. doi: 10.1016/s0168-8278(98)80224-9. PMID 9625309